CLINICAL TRIAL: NCT02961842
Title: Combined Colloid Preload And Crystalloid Coload Versus Crystalloid Coload During Spinal Anesthesia for Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Mohamed Tawfik, Lecturer, Department of anesthesia and surgical intensive care, principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R/16.09.64
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Anesthesia, Spinal; Cesarean Section
MeSH Terms: interventions — Anesthesia, Spinal; Cesarean Section

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination (Experimental): 500 mL colloid preload and 500 mL crystalloid coload. Cesarean delivery performed under spinal anesthesia (intrathecal bupivacaine 12.5 mg and intrathecal fentanyl 15 µg). Ultrasound assessment of the Inferior vena cava diameter. Intravenous ephedrine will be administered.
  Interventions: Drug: 500 mL Colloid Preload; Procedure: Spinal Anesthesia; Drug: Intrathecal Bupivacaine; Drug: Intrathecal Fentanyl; Drug: 500 mL Crystalloid Coload; Procedure: Cesarean Delivery; Radiation: Ultrasound Assessment of the Inferior Vena Cava; Drug: Intravenous Ephedrine
- Coload (Active Comparator): 1000 mL crystalloid coload. Cesarean delivery performed under spinal anesthesia (intrathecal bupivacaine 12.5 mg and intrathecal fentanyl 15 µg). Ultrasound assessment of the Inferior vena cava diameter. Intravenous ephedrine will be administered.
  Interventions: Procedure: Spinal Anesthesia; Drug: Intrathecal Bupivacaine; Drug: Intrathecal Fentanyl; Drug: 1000 mL Crystalloid Coload; Procedure: Cesarean Delivery; Radiation: Ultrasound Assessment of the Inferior Vena Cava; Drug: Intravenous Ephedrine

INTERVENTIONS:
Drug: 500 mL Colloid Preload — 6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride (voluven®) 500 mL will be rapidly infused before spinal anesthesia
  Arms: Combination
Procedure: Spinal Anesthesia — Performed at the L3-L4 or L4-L5 interspace using 27- or 25-gauge spinal needle
Drug: Intrathecal Bupivacaine — Bupivacaine 12.5 mg (2.5 mL 0.5%) will be administered in the subarachnoid space
Drug: Intrathecal Fentanyl — Fentanyl 15 µg will be administered in the subarachnoid space
Drug: 500 mL Crystalloid Coload — Ringer acetate 500 mL will be rapidly infused immediately after intrathecal injection
  Arms: Combination
Drug: 1000 mL Crystalloid Coload — Ringer acetate 1000 mL will be rapidly infused immediately after intrathecal injection
  Arms: Coload
Procedure: Cesarean Delivery — Lower segment cesarean section using the Pfannenstiel incision
Radiation: Ultrasound Assessment of the Inferior Vena Cava — The inferior vena cava largest and smallest diameters will be measured proximal to the opening of the hepatic veins in the longitudinal axis with the M-mode using a 5-2 MHz curved array ultrasound probe placed longitudinally in the subxiphoid region
Drug: Intravenous Ephedrine — Intravenous ephedrine 3, 5, and 10 mg will be administered when Systolic blood pressure decreases below 90%, 80%, and 70% of baseline, respectively.

SUMMARY:
The study will compare one technique of fluid administration (combined colloid preload and crystalloid colaod) with another one (crystalloid coload) during elective cesarean delivery performed under spinal anesthesia.

DETAILED DESCRIPTION:
This randomized, controlled, double-blind study will be conducted on ASA physical status II parturients with full-term singleton pregnancy undergoing elective cesarean delivery under spinal anesthesia. Participants will receive either 500 mL colloid preload and 500 mL crystalloid coload (Combination group) or 1000 mL crystalloid coload (Coload group). Systolic blood pressure will be recorded every minute and ephedrine will be administered when hypotension occurs according to a predefined protocol. The total ephedrine dose, time to the first ephedrine dose, heart rate, inferior vena cava diameter, nausea/vomiting, and neonatal Apgar scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status II parturients
* Full term, singleton pregnancy
* Elective cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Age <19 or > 40 years
* Height <150 cm
* Weight <60 kg
* Body mass index ≥40 kg/m2
* Contraindications to spinal anesthesia (increased intracranial pressure, coagulopathy, or local skin infection)
* Chronic or pregnancy-induced hypertension
* Hemoglobin <10 gm/dL.
* Diabetes mellitus, cardiovascular, cerebrovascular, or renal disease
* Polyhydramnios or known fetal abnormalities

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-11-20 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
Total ephedrine dose | intraoperative

SECONDARY OUTCOMES:
Incidence of hypotension | intraoperative
  Hypotension: Systolic blood pressure <80% of baseline
Incidence of severe hypotension | intraoperative
  Severe hypotension: Systolic blood pressure <70% of baseline
Time to the first ephedrine dose | intraoperative
Heart rate | intraoperative
Inferior vena cava largest and smallest diameters | Baseline, at 1 and 5 minutes after intrathecal injection, delivery
Inferior vena cava collapsibility index | Baseline, at 1 and 5 minutes after intrathecal injection, delivery
  Collapsibility index = (Largest diameter - Smallest diameter) / Largest diameter
Incidence of nausea and/or vomiting | intraoperative
Neonatal Apgar score | At 1 and 5 minutes after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Tawfik, MD, Principal Investigator — Mansoura University Hospital
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tawfik MM, Tarbay AI, Elaidy AM, Awad KA, Ezz HM, Tolba MA. Combined Colloid Preload and Crystalloid Coload Versus Crystalloid Coload During Spinal Anesthesia for Cesarean Delivery: A Randomized Controlled Trial. Anesth Analg. 2019 Feb;128(2):304-312. doi: 10.1213/ANE.0000000000003306. PMID 29461392